CLINICAL TRIAL: NCT01311661
Title: Phase II, Randomised, Double-Blind, Cross-over Study to Compare the 24-hour FEV1-time Profile of Orally Inhaled Olodaterol, Delivered With the Respimat® Inhaler, After 3 Weeks of Olodaterol Once Daily Medium Dose, Twice Daily Low Dose and Placebo or After 3 Weeks of Once Daily High Dose, Twice Daily Medium Dose and Placebo Administration in Patients With Moderate to Severe Persistent Asthma
Brief Title: A Study to Compare the Efficacy and Safety of Different Dosings of Olodaterol Administered With the Respimat® Inhaler in Patients With Moderate to Severe Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1222.29; 2008-006625-14 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-03-04; First posted 2011-03-09 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

ARMS (2):
- Olodaterol medium daily dose (Experimental): Olodaterol medium daily dose given either as once daily or split into two low doses daily or placebo only in randomised sequence of three cross-over treatment phases
  Interventions: Drug: Olodaterol low daily dose twice daily; Drug: Placebo twice daily; Drug: Olodaterol medium daily dose once daily and placebo
- Olodaterol high daily dose (Experimental): Olodaterol high daily dose given either as once daily or split into two medium doses daily or placebo only in randomised sequence of three cross-over treatment phases
  Interventions: Drug: Placebo twice daily; Drug: Olodaterol medium daily dose twice daily; Drug: Olodaterol high daily dose once daily and placebo

INTERVENTIONS:
Drug: Placebo twice daily — Inhaled Placebo of Olodaterol twice daily
  Arms: Olodaterol high daily dose
Drug: Olodaterol low daily dose twice daily — Inhaled Olodaterol medium daily dose administered as low dose twice daily
  Arms: Olodaterol medium daily dose
Drug: Olodaterol medium daily dose twice daily — Inhaled Olodaterol high daily dose administered as medium dose twice daily
  Arms: Olodaterol high daily dose
Drug: Placebo twice daily — Inhaled Placebo of Olodaterol twice daily
  Arms: Olodaterol medium daily dose
Drug: Olodaterol high daily dose once daily and placebo — Inhaled Olodaterol high daily dose administered as one full dose once daily and placebo once daily
  Arms: Olodaterol high daily dose
Drug: Olodaterol medium daily dose once daily and placebo — Inhaled Olodaterol medium daily dose administered as one full dose once daily and placebo once daily
  Arms: Olodaterol medium daily dose

SUMMARY:
This study will compare efficacy and safety of different regimens of olodaterol administration in asthma (once daily, twice daily) with placebo in a complete cross-over design each within one of the two daily dose groups (medium or high daily dose).

ELIGIBILITY:
Inclusion criteria:

1. Patients of either sex.
2. Aged 18 to 70 years.
3. A current diagnosis and a documented minimum 3 month history of asthma Global Initiative for Asthma (GINA) treatment steps 3 and 4.
4. Prebronchodilator Forced Expiratory Volume in one second (FEV1) >= 60% predicted and < 90% predicted according to European Coal and Steel Community (ECSC).
5. Increase in FEV1 >=12% and >=200 mL 15 min. after 400 µg salbutamol (albuterol);
6. Stable on medium to high dose inhaled corticosteroids (ICS) or low to high dose ICS in combination with a long acting beta-adrenergics (LABA) for at least 6 weeks prior to screening. Stable on ICS mono component of the former fixed LABA/ICS treatment for at least 48 hours prior to Visit 1b.

Exclusion criteria:

1. Patients with a significant disease other than asthma.
2. History of frequent seasonal exacerbations of asthma (defined as one or more seasonal exacerbations every year for the past three years).
3. Upper respiratory tract infection in the past 3 weeks prior to screening visit 1b.
4. Oral or other systemic corticosteroids in the past 6 weeks.
5. Patients with allergen desensitization therapy if started within two years, if they are not on an established maintenance regimen characterized by dose adjustments but no further increase to the tolerable maximum in the same course of immunotherapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (36):
- United States (12):
  - 1222.29.11006 Boehringer Ingelheim Investigational Site, Huntington Beach, California
  - 1222.29.11001 Boehringer Ingelheim Investigational Site, Centennial, Colorado
  - 1222.29.11012 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 1222.29.11002 Boehringer Ingelheim Investigational Site, Overland Park, Kansas
  - 1222.29.11004 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 1222.29.11011 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1222.29.11009 Boehringer Ingelheim Investigational Site, Skillman, New Jersey
  - 1222.29.11003 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 1222.29.11008 Boehringer Ingelheim Investigational Site, Canton, Ohio
  - 1222.29.11007 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1222.29.11005 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1222.29.11010 Boehringer Ingelheim Investigational Site, Richmond, Virginia
- Austria (4):
  - 1222.29.43003 Boehringer Ingelheim Investigational Site, Linz
  - 1222.29.43002 Boehringer Ingelheim Investigational Site, Schlüsslberg
  - 1222.29.43001 Boehringer Ingelheim Investigational Site, Thalheim bei Wels
  - 1222.29.43004 Boehringer Ingelheim Investigational Site, Wels
- Germany (10):
  - 1222.29.49004 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.29.49006 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.29.49007 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.29.49008 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.29.49002 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1222.29.49010 Boehringer Ingelheim Investigational Site, Großhansdorf
  - 1222.29.49003 Boehringer Ingelheim Investigational Site, Lübeck
  - 1222.29.49005 Boehringer Ingelheim Investigational Site, Rüdersdorf
  - 1222.29.49001 Boehringer Ingelheim Investigational Site, Wiesbaden
  - 1222.29.49009 Boehringer Ingelheim Investigational Site, Wiesloch
- Hungary (4):
  - 1222.29.36002 Boehringer Ingelheim Investigational Site, Mosonmagyaróvár
  - 1222.29.36003 Boehringer Ingelheim Investigational Site, Nyíregyháza
  - 1222.29.36001 Boehringer Ingelheim Investigational Site, Sopron
  - 1222.29.36004 Boehringer Ingelheim Investigational Site, Zalaegerszeg
- Slovakia (4):
  - 1222.29.42001 Boehringer Ingelheim Investigational Site, Bardejov
  - 1222.29.42002 Boehringer Ingelheim Investigational Site, Martin
  - 1222.29.42004 Boehringer Ingelheim Investigational Site, Nitra
  - 1222.29.42003 Boehringer Ingelheim Investigational Site, Spišská Nová Ves
- Slovenia (2):
  - 1222.29.38003 Boehringer Ingelheim Investigational Site, Golnik
  - 1222.29.38002 Boehringer Ingelheim Investigational Site, Kamnik

REFERENCES:
- [Derived] Beeh KM, LaForce C, Gahlemann M, Wenz A, Toorawa R, Flezar M. Randomised, double-blind, placebo-controlled crossover study to investigate different dosing regimens of olodaterol delivered via Respimat(R) in patients with moderate to severe persistent asthma. Respir Res. 2015 Jul 16;16(1):87. doi: 10.1186/s12931-015-0243-1. PMID 26177937

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Total: This was a double-blind, 3-period crossover trial. 206 patients were assigned randomly to one of 12 treatment sequences with either 5 microgram (mcg) Olodaterol (Olo) once daily (qd) and 2.5 mcg Olodaterol twice daily (bid) and placebo (6 sequences) or 10 mcg Olodaterol qd and 5 mcg Olodaterol bid and placebo (6 sequences). The duration of each treatment period was 3 weeks separated by washout periods of 2 weeks.
Period: Overall Study
Arm/Group | Study Total
Started | 206 (Entered and treated)
Received Placebo | 201
Received Olo 2.5 mcg Bid | 101
Received Olo 5 mcg qd | 101
Received Olo 5 mcg Bid | 101
Received Olo 10 mcg qd | 102
Completed | 199
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Study Total
Number analyzed (Participants) | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109
  Male | 97

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-24 Hours (AUC 0-24h) Response at the End of Each Treatment Period
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values at the randomisation visit. Means are adjusted for treatment, period, patient and study baseline. FEV1 AUC 0-24h was calculated from 0-24 hours post-dose using the trapezoidal rule, divided by the observation time (24h) to report in litres.
Time Frame: 1 hour (h) prior and 10 minutes (min) prior to first dose (baseline) and -1 h, -10 mins, 30 min, 60 min, 2 h, 3 h, 4 h, 6 h, 8 h, 10 h, 11 h 50 min, 12 h 30 min, 13 h, 14 h, 22 h, 23 h, and 23 h 50 min related to morning dose after 3 weeks
Population: Full analysis set (FAS). FAS is defined as all patients in the treated set for whom the baseline (pre-dose) value is available, and who have a value for the primary endpoint for at least one crossover period.
Measure: Mean (Standard Error); unit: Liter
Groups:
- Placebo: Matching Placebo delivered by the Respimat Inhaler. Two actuations bid (morning and evening dosing).
- Olo 2.5 mcg Bid: Olodaterol 2.5 mcg bid delivered by the Respimat Inhaler.
- Olo 5 mcg qd: Olodaterol 5 mcg qd (morning) and matching Placebo in the evening delivered by the Respimat Inhaler.
- Olo 5 mcg Bid: Olodaterol 5 mcg bid delivered by the Respimat Inhaler.
- Olo 10 mcg qd: Olodaterol 10 mcg qd (morning) and matching Placebo in the evening delivered by the Respimat Inhaler.
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 99 | 99 | 100 | 101
Liter | 0.022 (0.020) | 0.213 (0.024) | 0.173 (0.024) | 0.250 (0.024) | 0.231 (0.024)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted using a mixed model with treatment, period and study baseline value as fixed effects; and patients as random effect; Mean Difference (Final Values) = 0.191, 95% CI [0.152 to 0.229], Standard Error of Mean 0.020 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.150, 95% CI [0.111 to 0.189], Standard Error of Mean 0.020 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.228, 95% CI [0.190 to 0.266], Standard Error of Mean 0.020 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.209, 95% CI [0.170 to 0.247], Standard Error of Mean 0.020 — Olo 10 mcg qd minus Placebo

2. Secondary Outcome: FEV1 Area Under Curve 0-12 Hours (AUC 0-12h) Response at the End of Each Treatment Period
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values at the randomisation visit. Means are adjusted for treatment, period, patient and study baseline. FEV1 AUC 0-12h was calculated from 0-12 hours post-dose using the trapezoidal rule, divided by the observation time (12h) to report in litres.
Time Frame: 1 hour (h) prior and 10 minutes (min) prior to first dose (baseline) and -1 h, -10 mins, 30 min, 60 min, 2 h, 3 h, 4 h, 6 h, 8 h, 10 h, 11 h 50 min related to morning dose after 3 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 99 | 99 | 100 | 101
Liter | 0.052 (0.020) | 0.242 (0.024) | 0.212 (0.024) | 0.266 (0.024) | 0.272 (0.024)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.190, 95% CI [0.150 to 0.229], Standard Error of Mean 0.020 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.160, 95% CI [0.121 to 0.199], Standard Error of Mean 0.020 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.214, 95% CI [0.175 to 0.253], Standard Error of Mean 0.020 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.219, 95% CI [0.181 to 0.258], Standard Error of Mean 0.020 — Olo 10 mcg qd minus Placebo

3. Secondary Outcome: FEV1 Area Under Curve 12-24 Hours (AUC 12-24h) Response at the End of Each Treatment Period
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values at the randomisation visit. Means are adjusted for treatment, period, patient and study baseline. FEV1 AUC 12-24h was calculated from 12-24 hours post-dose using the trapezoidal rule, divided by the observation time (12h) to report in litres.
Time Frame: 1 hour (h) prior and 10 minutes (min) prior to first dose (baseline) and 11 h 50 min, 12 h 30 min, 13 h, 14 h, 22 h, 23 h, and 23 h 50 min related to morning dose after 3 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 201 | 99 | 99 | 100 | 101
Liter | -0.010 (0.020) | 0.186 (0.025) | 0.135 (0.025) | 0.233 (0.025) | 0.189 (0.025)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.196, 95% CI [0.153 to 0.238], Standard Error of Mean 0.022 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.144, 95% CI [0.102 to 0.187], Standard Error of Mean 0.022 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.242, 95% CI [0.200 to 0.285], Standard Error of Mean 0.022 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.198, 95% CI [0.156 to 0.241], Standard Error of Mean 0.022 — Olo 10 mcg qd minus Placebo

4. Secondary Outcome: Peak FEV1 Within 24 Hours Post-dose Response
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values at the randomisation visit. Peak FEV1 within 24 hours post dose measured following the morning trial drug inhalation at the end of each 3 week period of randomised treatment. Means are adjusted for treatment, period, patient and study baseline.
Time Frame: 1 hour (h) prior and 10 minutes (min) prior to first dose (baseline) and 30 min, 60 min, 2 h, 3 h, 4 h, 6 h, 8h, 10 h, 11 h 50 min, 12 h 30 min, 13 h, 14 h, 22 h, 23 h, and 23 h 50 min related to morning dose after 3 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 201 | 99 | 99 | 100 | 101
Liter | 0.227 (0.021) | 0.410 (0.027) | 0.380 (0.027) | 0.449 (0.027) | 0.437 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.183, 95% CI [0.138 to 0.228], Standard Error of Mean 0.023 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.153, 95% CI [0.108 to 0.198], Standard Error of Mean 0.023 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.222, 95% CI [0.177 to 0.267], Standard Error of Mean 0.023 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.210, 95% CI [0.165 to 0.255], Standard Error of Mean 0.023 — Olo 10 mcg qd minus Placebo

5. Secondary Outcome: Trough FEV1 Response
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values at the randomisation visit. Trough values were defined as the mean of 2 FEV1 values performed at 23 h and 23 h 50 min after the last morning trial drug inhalation at the end of each 3 week period of randomised treatment. Means are adjusted for treatment, period, patient and study baseline.
Time Frame: 1 hour (h) prior and 10 minutes (min) prior to first dose (baseline) and 23 h, and 23 h 50 min related to morning dose after 3 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 201 | 99 | 99 | 100 | 101
Liter | 0.033 (0.022) | 0.189 (0.027) | 0.134 (0.027) | 0.229 (0.027) | 0.205 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.156, 95% CI [0.109 to 0.203], Standard Error of Mean 0.024 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.101, 95% CI [0.054 to 0.148], Standard Error of Mean 0.024 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.196, 95% CI [0.149 to 0.243], Standard Error of Mean 0.024 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.172, 95% CI [0.125 to 0.219], Standard Error of Mean 0.024 — Olo 10 mcg qd minus Placebo

6. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-12 Hours (AUC 0-12h) Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values at the randomisation visit. Means are adjusted for treatment, period, patient and study baseline. FVC AUC 0-12h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: as for outcome 2
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 99 | 99 | 100 | 101
Liter | -0.004 (0.022) | 0.132 (0.027) | 0.119 (0.027) | 0.138 (0.026) | 0.143 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.136, 95% CI [0.091 to 0.180], Standard Error of Mean 0.023 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.122, 95% CI [0.078 to 0.167], Standard Error of Mean 0.023 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.142, 95% CI [0.098 to 0.186], Standard Error of Mean 0.022 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.147, 95% CI [0.103 to 0.191], Standard Error of Mean 0.022 — Olo 10 mcg qd minus Placebo

7. Secondary Outcome: FVC Area Under Curve 12-24 Hours (AUC 12-24h) Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values at the randomisation visit. Means are adjusted for treatment, period, patient and study baseline. FVC AUC 12-24h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: as for outcome 3
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 201 | 99 | 99 | 100 | 101
Liter | -0.056 (0.023) | 0.102 (0.028) | 0.081 (0.028) | 0.114 (0.028) | 0.079 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.158, 95% CI [0.110 to 0.206], Standard Error of Mean 0.024 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.137, 95% CI [0.090 to 0.185], Standard Error of Mean 0.024 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.170, 95% CI [0.123 to 0.218], Standard Error of Mean 0.024 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.135, 95% CI [0.087 to 0.182], Standard Error of Mean 0.024 — Olo 10 mcg qd minus Placebo

8. Secondary Outcome: FVC Area Under Curve 0-24 Hours (AUC 0-24h) Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values at the randomisation visit. Means are adjusted for treatment, period, patient and study baseline. FVC AUC 0-24h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: 1 hour (h) prior and 10 minutes (min) prior to first dose (baseline) and -1 h, -10 mins, 30 min, 60 min, 2 h, 3 h, 4 h, 6 h, 8h, 10 h, 11 h 50 min, 12 h 30 min, 13 h, 14 h, 22 h, 23 h, and 23 h 50 min related to morning dose after 3 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 99 | 99 | 100 | 101
Liter | -0.029 (0.021) | 0.116 (0.026) | 0.099 (0.026) | 0.127 (0.026) | 0.111 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.145, 95% CI [0.102 to 0.188], Standard Error of Mean 0.022 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.128, 95% CI [0.085 to 0.171], Standard Error of Mean 0.022 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.156, 95% CI [0.113 to 0.198], Standard Error of Mean 0.022 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.140, 95% CI [0.098 to 0.182], Standard Error of Mean 0.022 — Olo 10 mcg qd minus Placebo

9. Secondary Outcome: Peak FVC Within 24 Hours Post-dose Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values at the randomisation visit. Peak FVC within 24 hours post-dose measured following the morning trial drug inhalation at the end of each 3 week period of randomised treatment. Means are adjusted for treatment, period, patient and study baseline.
Time Frame: as for outcome 4
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 201 | 99 | 99 | 100 | 101
Liter | 0.246 (0.024) | 0.382 (0.030) | 0.371 (0.030) | 0.390 (0.030) | 0.373 (0.029)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.136, 95% CI [0.084 to 0.187], Standard Error of Mean 0.026 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.124, 95% CI [0.073 to 0.176], Standard Error of Mean 0.026 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.144, 95% CI [0.093 to 0.195], Standard Error of Mean 0.026 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.126, 95% CI [0.075 to 0.177], Standard Error of Mean 0.026 — Olo 10 mcg qd minus Placebo

10. Secondary Outcome: Trough FVC Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values at the randomisation visit. Trough values were defined as the mean of 2 FVC values performed at 23 h and 23 h 50 min after the last morning trial drug inhalation at the end of each 3 week period of randomised treatment. Means are adjusted for treatment, period, patient and study baseline.
Time Frame: as for outcome 5
Population: FAS
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 201 | 99 | 99 | 100 | 101
Liter | -0.013 (0.024) | 0.096 (0.031) | 0.079 (0.031) | 0.105 (0.031) | 0.098 (0.031)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.110, 95% CI [0.055 to 0.165], Standard Error of Mean 0.028 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0010, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.092, 95% CI [0.037 to 0.147], Standard Error of Mean 0.028 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.118, 95% CI [0.063 to 0.172], Standard Error of Mean 0.028 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.111, 95% CI [0.057 to 0.166], Standard Error of Mean 0.028 — Olo 10 mcg qd minus Placebo

11. Secondary Outcome: Peak Expiratory Flow (PEF) Area Under Curve 0-12 Hours (AUC 0-12h) Response
Description: Response was defined as change from baseline. Study baseline PEF was defined as the mean of the available pre-dose PEF values at the randomisation visit. Means are adjusted for treatment, period, patient and study baseline. PEF AUC 0-12h was calculated using the trapezoidal rule, divided by the observation time to report in litres/seconds.
Time Frame: 1 hour (h) prior and 10 minutes (min) prior to first dose (baseline) and -1 h, -10 mins, 30 min, 60 min, 2 h, 3 h, 4 h, 6 h, 8h, 10 h, 11 h 50 min related to morning dose after 3 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter/sec
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 99 | 99 | 100 | 101
Liter/sec | 0.101 (0.060) | 0.730 (0.075) | 0.703 (0.075) | 0.732 (0.074) | 0.787 (0.074)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.629, 95% CI [0.500 to 0.757], Standard Error of Mean 0.065 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.601, 95% CI [0.473 to 0.730], Standard Error of Mean 0.065 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.631, 95% CI [0.503 to 0.758], Standard Error of Mean 0.065 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.685, 95% CI [0.558 to 0.813], Standard Error of Mean 0.065 — Olo 10 mcg qd minus Placebo

12. Secondary Outcome: PEF Area Under Curve 12-24 Hours (AUC 12-24h) Response
Description: Response was defined as change from baseline. Study baseline PEF was defined as the mean of the available pre-dose PEF values at the randomisation visit. Means are adjusted for treatment, period, patient and study baseline. PEF AUC 12-24h was calculated using the trapezoidal rule, divided by the observation time to report in litres/seconds.
Time Frame: as for outcome 3
Population: FAS
Measure: Mean (Standard Error); unit: Liter/sec
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 201 | 99 | 99 | 100 | 101
Liter/sec | -0.135 (0.061) | 0.530 (0.077) | 0.430 (0.076) | 0.567 (0.076) | 0.464 (0.076)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.665, 95% CI [0.532 to 0.799], Standard Error of Mean 0.068 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.564, 95% CI [0.431 to 0.698], Standard Error of Mean 0.068 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.702, 95% CI [0.569 to 0.835], Standard Error of Mean 0.068 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.599, 95% CI [0.467 to 0.732], Standard Error of Mean 0.067 — Olo 10 mcg qd minus Placebo

13. Secondary Outcome: Peak Expiratory Flow (PEF) Area Under Curve 0-24 Hours (AUC 0-24h) Response
Description: Response was defined as change from baseline. Study baseline PEF was defined as the mean of the available pre-dose PEF values at the randomisation visit. Means are adjusted for treatment, period, patient and study baseline. PEF AUC 0-24h was calculated using the trapezoidal rule, divided by the observation time to report in litres/seconds.
Time Frame: as for outcome 8
Population: FAS
Measure: Mean (Standard Error); unit: Liter/sec
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 200 | 99 | 99 | 100 | 101
Liter/sec | -0.014 (0.059) | 0.627 (0.073) | 0.563 (0.073) | 0.653 (0.073) | 0.629 (0.073)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.641, 95% CI [0.516 to 0.765], Standard Error of Mean 0.063 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.577, 95% CI [0.453 to 0.701], Standard Error of Mean 0.063 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.667, 95% CI [0.544 to 0.790], Standard Error of Mean 0.063 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.643, 95% CI [0.519 to 0.766], Standard Error of Mean 0.063 — Olo 10 mcg qd minus Placebo

14. Secondary Outcome: Peak PEF Within 24 Hours Post-dose Response
Description: Response was defined as change from baseline. Study baseline PEF was defined as the mean of the available pre-dose PEF values at the randomisation visit. Peak PEF within 24 hours post dose measured following the morning trial drug inhalation at the end of each 3 week period of randomised treatment. Means are adjusted for treatment, period, patient and study baseline.
Time Frame: as for outcome 4
Population: FAS
Measure: Mean (Standard Error); unit: Liter/sec
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 201 | 99 | 99 | 100 | 101
Liter/sec | 0.663 (0.068) | 1.254 (0.087) | 1.185 (0.087) | 1.257 (0.086) | 1.286 (0.086)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.591, 95% CI [0.436 to 0.746], Standard Error of Mean 0.079 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.522, 95% CI [0.366 to 0.677], Standard Error of Mean 0.079 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.594, 95% CI [0.439 to 0.749], Standard Error of Mean 0.079 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.623, 95% CI [0.468 to 0.777], Standard Error of Mean 0.079 — Olo 10 mcg qd minus Placebo

15. Secondary Outcome: Trough PEF Response
Description: Response was defined as change from baseline. Study baseline PEF was defined as the mean of the available pre-dose PEF values at the randomisation visit. Trough values were defined as the mean of 2 PEF values performed at 23 h and 23 h 50 min after the last morning trial drug inhalation at the end of each 3 week period of randomised treatment. Means are adjusted for treatment, period, patient and study baseline.
Time Frame: as for outcome 5
Population: FAS
Measure: Mean (Standard Error); unit: Liter/sec
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 201 | 99 | 99 | 100 | 101
Liter/sec | -0.009 (0.062) | 0.520 (0.078) | 0.401 (0.078) | 0.594 (0.077) | 0.472 (0.077)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.529, 95% CI [0.396 to 0.662], Standard Error of Mean 0.068 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.410, 95% CI [0.277 to 0.543], Standard Error of Mean 0.068 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.603, 95% CI [0.471 to 0.736], Standard Error of Mean 0.067 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.481, 95% CI [0.349 to 0.613], Standard Error of Mean 0.067 — Olo 10 mcg qd minus Placebo

16. Secondary Outcome: Mean Pre-dose Morning PEF (PEF a.m.)
Description: PEF a.m. was measured by patients at home using the AM3 device (overall means obtained during each period of randomised treatment will be compared). Means are adjusted for treatment, period, patient and study baseline.
Time Frame: 0-3 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter/min
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 201 | 99 | 100 | 101 | 101
Liter/min | 395.36 (2.857) | 428.32 (3.586) | 427.99 (3.575) | 427.02 (3.562) | 424.26 (3.562)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 32.957, 95% CI [26.709 to 39.206], Standard Error of Mean 3.180 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 32.632, 95% CI [26.409 to 38.855], Standard Error of Mean 3.167 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 31.660, 95% CI [25.448 to 37.872], Standard Error of Mean 3.161 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 28.895, 95% CI [22.683 to 35.107], Standard Error of Mean 3.161 — Olo 10 mcg qd minus Placebo

17. Secondary Outcome: Mean Pre-dose Evening PEF (PEF p.m.)
Description: PEF p.m. was measured by patients at home using the AM3 device (overall means obtained during each period of randomised treatment will be compared). Means are adjusted for treatment, period, patient and study baseline.
Time Frame: 0-3 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Liter/min
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 201 | 99 | 100 | 101 | 101
Liter/min | 409.93 (2.717) | 438.80 (3.418) | 441.98 (3.407) | 441.74 (3.395) | 443.25 (3.395)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 28.870, 95% CI [22.884 to 34.856], Standard Error of Mean 3.046 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 32.056, 95% CI [26.094 to 38.018], Standard Error of Mean 3.034 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 31.816, 95% CI [25.864 to 37.767], Standard Error of Mean 3.028 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 33.327, 95% CI [27.375 to 39.278], Standard Error of Mean 3.028 — Olo 10 mcg qd minus Placebo

18. Secondary Outcome: PEF Daily Variability
Description: PEF daily variability was assessed by patients at home using the AM3 device (overall means obtained during each period of randomised treatment will be compared). PEF daily variability is the absolute difference between the morning and the evening PEF value divided by the mean of these two values, expressed as a percent. Means are adjusted for treatment, period, patient and study baseline.
Time Frame: 0-3 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 201 | 99 | 100 | 101 | 101
Percentage | 10.157 (0.288) | 8.576 (0.371) | 8.732 (0.369) | 8.419 (0.368) | 9.468 (0.368)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.581, 95% CI [-2.262 to -0.900], Standard Error of Mean 0.346 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.426, 95% CI [-2.104 to -0.748], Standard Error of Mean 0.345 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.738, 95% CI [-2.415 to -1.062], Standard Error of Mean 0.344 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0458, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.689, 95% CI [-1.366 to -0.013], Standard Error of Mean 0.344 — Olo 10 mcg qd minus Placebo

19. Secondary Outcome: Mean Pre-dose Morning FEV1 (FEV1 a.m.)
Description: FEV1 a.m. was measured by patients at home using the AM3 device (overall means obtained during each period of randomised treatment will be compared). Means are adjusted for treatment, period, patient and study baseline.
Time Frame: 0-3 weeks
Population: FAS
Measure: Mean (Standard Error); unit: mL
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 201 | 99 | 100 | 101 | 101
mL | 2425.1 (17.870) | 2598.5 (22.276) | 2580.2 (22.208) | 2574.3 (22.133) | 2575.5 (22.133)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 173.391, 95% CI [135.099 to 211.682], Standard Error of Mean 19.484 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 155.097, 95% CI [116.961 to 193.234], Standard Error of Mean 19.406 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 149.268, 95% CI [111.204 to 187.333], Standard Error of Mean 19.369 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 150.441, 95% CI [112.377 to 188.505], Standard Error of Mean 19.369 — Olo 10 mcg qd minus Placebo

20. Secondary Outcome: Mean Pre-dose Evening FEV1 (FEV1 p.m.)
Description: FEV1 p.m. was measured by patients at home using the AM3 device (overall means obtained during each period of randomised treatment will be compared). Means are adjusted for treatment, period, patient and study baseline.
Time Frame: 0-3 weeks
Population: FAS
Measure: Mean (Standard Error); unit: mL
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 201 | 99 | 100 | 101 | 101
mL | 2474.3 (17.692) | 2616.6 (21.949) | 2606.5 (21.884) | 2616.5 (21.810) | 2631.7 (21.809)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 142.251, 95% CI [104.916 to 179.586], Standard Error of Mean 18.997 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 132.138, 95% CI [94.954 to 169.322], Standard Error of Mean 18.920 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 142.136, 95% CI [105.021 to 179.251], Standard Error of Mean 18.885 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 157.306, 95% CI [120.192 to 194.420], Standard Error of Mean 18.885 — Olo 10 mcg qd minus Placebo

21. Secondary Outcome: Mean Number of Puffs of Rescue Medication During the Whole Day
Description: Mean of daily use of salbutamol (albuterol) rescue medication as needed during the entire study period. Assessed by patients at home using the AM3 device (overall mean number obtained during each period of randomised treatment will be compared). Means are adjusted for treatment, period, patient and study baseline.
Time Frame: 0-3 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Puffs
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 201 | 99 | 100 | 101 | 101
Puffs | 1.665 (0.091) | 1.110 (0.120) | 1.028 (0.119) | 1.077 (0.119) | 1.119 (0.119)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.554, 95% CI [-0.780 to -0.329], Standard Error of Mean 0.115 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.637, 95% CI [-0.862 to -0.412], Standard Error of Mean 0.114 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.588, 95% CI [-0.813 to -0.364], Standard Error of Mean 0.114 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.546, 95% CI [-0.770 to -0.322], Standard Error of Mean 0.114 — Olo 10 mcg qd minus Placebo

22. Secondary Outcome: Percentage of Asthma Symptom Free Days
Description: Percentage of asthma-symptom free days of each treatment period was calculated as the number of symptom-free days divided by the number of days on treatment multiplied by 100. A symptom-free day was defined as a day in which no asthma symptoms were recorded, no rescue medication was recorded, activities during the day were not at all limited due to asthma, no shortness of breath during the day was recorded, no wheezing or coughing during the day and no night-time awakenings due to asthma were recorded. Assessed by patients at home using the AM3 device.
Time Frame: 0-3 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Percentage of asthma symptom free days
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 201 | 99 | 100 | 101 | 101
Percentage of asthma symptom free days | 23.630 (2.235) | 33.929 (3.554) | 36.306 (3.644) | 28.844 (3.271) | 28.049 (3.368)

23. Secondary Outcome: Number of Patients Categorized by Highest Number of Night Time Awakenings (Overall)
Description: Assessed by patients at home using the AM3 device during each period of randomised treatment.
Time Frame: 0-3 weeks
Population: FAS
Measure: Number; unit: Number of patients
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 201 | 99 | 100 | 101 | 101
Number of patients
  Did not wake up | 93 | 50 | 53 | 44 | 47
  Woke up once | 67 | 31 | 36 | 41 | 32
  Woke up 2-5 times | 36 | 18 | 10 | 14 | 19
  Woke up > 5 times | 5 | 0 | 1 | 0 | 2
  Was awake all night | 0 | 0 | 0 | 2 | 1

24. Secondary Outcome: Number of Patients Categorized by Worst Asthma Daytime Symptoms (Overall)
Description: Assessed by patients at home using the AM3 device during each period of randomised treatment .
Time Frame: 0-3 weeks
Population: FAS
Measure: Number; unit: Number of patients
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 201 | 99 | 100 | 101 | 101
Number of patients
  No asthma symptoms | 31 | 24 | 27 | 18 | 20
  Mild asthma symptoms | 66 | 45 | 42 | 42 | 41
  Moderate asthma symptoms | 85 | 25 | 27 | 36 | 37
  Severe asthma symptoms | 18 | 4 | 3 | 4 | 2
  Very severe asthma symptoms | 1 | 1 | 1 | 1 | 1

25. Secondary Outcome: Number of Patients Categorized by Worst Asthma Nighttime Symptoms (Overall)
Description: Assessed by patients at home using the AM3 device during each period of randomised treatment.
Time Frame: 0-3 weeks
Population: FAS
Measure: Number; unit: Number of patients
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 201 | 99 | 100 | 101 | 101
Number of patients
  No asthma symptoms | 39 | 32 | 29 | 21 | 21
  Mild asthma symptoms | 76 | 35 | 38 | 48 | 40
  Moderate asthma symptoms | 74 | 26 | 32 | 29 | 35
  Severe asthma symptoms | 9 | 4 | 1 | 2 | 3
  Very severe asthma symptoms | 3 | 2 | 0 | 1 | 2

26. Secondary Outcome: Total Asthma Control Questionnaire (ACQ) Score
Description: Control of asthma as assessed by the ACQ at the end of each 3-week treatment period.The ACQ contains 7 questions, each question has a 7 point scale from 0 (no symptoms) till 6 (highest intensity). Total score was defined as the sum of all items divided by the number of items.
Time Frame: 3 weeks
Population: FAS
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 201 | 99 | 100 | 101 | 101
Units on a scale | 1.613 (0.040) | 1.256 (0.053) | 1.317 (0.053) | 1.312 (0.053) | 1.311 (0.053)
Statistical Analysis 1: Comparison: Placebo vs Olo 2.5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.357, 95% CI [-0.461 to -0.253], Standard Error of Mean 0.053 — Olo 2.5 mcg bid minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.296, 95% CI [-0.400 to -0.192], Standard Error of Mean 0.053 — Olo 5 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olo 5 mcg Bid; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.301, 95% CI [-0.405 to -0.198], Standard Error of Mean 0.053 — Olo 5 mcg bid minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.302, 95% CI [-0.405 to -0.198], Standard Error of Mean 0.053 — Olo 10 mcg qd minus Placebo

27. Secondary Outcome: Clinical Relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis and ECG
Description: Clinical relevant abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis and ECG. New abnormal findings or worsening of baseline conditions were reported as Adverse Events. Time frame for adverse event reporting includes 12 days into the subsequent washout or post-treatment period.
Time Frame: 3 weeks + 12 days
Population: Treated set
Measure: Number; unit: Participants
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Number analyzed (Participants) | 201 | 101 | 101 | 101 | 102
Participants
  Atrioventricular block first degree | 0 | 0 | 1 | 0 | 0
  Sinus tachycardia | 1 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased | 0 | 0 | 0 | 0 | 1
  Blood creatinine increased | 0 | 0 | 1 | 0 | 0
  Blood glucose increased | 0 | 0 | 0 | 0 | 1
  Blood urea abnormal | 0 | 0 | 1 | 0 | 0
  Gamma-glutamyltransferase increased | 0 | 0 | 0 | 0 | 1
  Blood creatine phosphokinase increased | 1 | 0 | 0 | 0 | 0
  Blood urine present | 1 | 0 | 0 | 0 | 0
  Anaemia | 0 | 0 | 0 | 1 | 0
  Hypertension | 0 | 0 | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: 3 weeks treatment period + 12 days
Description: Time frame for adverse event reporting includes 12 days into the subsequent washout or post-treatment period.
Arm/Group | Placebo | Olo 2.5 mcg Bid | Olo 5 mcg qd | Olo 5 mcg Bid | Olo 10 mcg qd
Serious Adverse Events (participants affected / at risk) | 2/201 | 1/101 | 0/101 | 1/101 | 0/102
Other Adverse Events (participants affected / at risk) | 0/201 | 0/101 | 0/101 | 0/101 | 0/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=201) | Olo 2.5 mcg Bid (N=101) | Olo 5 mcg qd (N=101) | Olo 5 mcg Bid (N=101) | Olo 10 mcg qd (N=102)
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication